CLINICAL TRIAL: NCT00003087
Title: Phase II Trial of Preoperative Combined Modality Therapy for Localized Esophageal Carcinoma: Cisplatin-Paclitaxel Followed by Radiation Therapy With Concurrent Cisplatin and Paclitaxel
Brief Title: Combination Chemotherapy, Radiation Therapy and Surgery in Treating Patients With Cancer of the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-088; CDR0000065787 (Registry Identifier: PDQ (Physician Data Query)); NCI-T97-0066
Record Dates: First submitted 1999-11-01; First posted 2004-08-02 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Paclitaxel; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: paclitaxel
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug with radiation therapy before surgery may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, radiation therapy, and surgery in treating patients with cancer of the esophagus that can be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate to preoperative induction paclitaxel/cisplatin followed by concurrent paclitaxel/cisplatin and radiotherapy in locally advanced esophageal cancer. II. Determine the toxic effects, including surgical morbidity and mortality, and patient survival after this combination therapy. III. Monitor the quality of life of patients receiving this combination therapy. IV. Determine c Jun oncogene and thymidylate synthase expression and p53 mutation before and after this combination therapy.

OUTLINE: This is an open label, multicenter study. (Adenocarcinoma stratum closed) Patients receive of induction chemotherapy consisting of paclitaxel IV over 3 hours followed by cisplatin IV on days 1 and 22. Patients then receive radiation therapy 5 days a week for 6 weeks, along with paclitaxel and cisplatin 4 days a week. Patients undergo surgery (complete or partial resection) within 4-8 weeks of completion of the chemoradiotherapy. Patients are followed every 3 months for the first 2 years, every 6 months for the next 2 years, and annually thereafter. Quality of life is assessed for the first year of follow up only.

PROJECTED ACCRUAL: A maximum of 25 patients will be accrued for each histology (adenocarcinoma, squamous carcinoma) within 18-24 months. (Adenocarcinoma stratum closed)

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (adenocarcinoma stratum closed) Locally advanced and surgically resectable (T2-4 N0-1 M0) T1 N1 tumors are eligible, T1 N0 tumors and in situ carcinoma are not eligible No cervical esophageal tumors No brain, pulmonary, liver, bone, lymph node (cervical or supraclavicular) or other distant metastases No positive cytology of the pleura, pericardium, or peritoneum No invasion of the tracheobronchial tree or presence of tracheoesophageal fistula

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1500/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Calcium no greater than 12 mg/dL Cardiovascular: No New York Heart Association class III/IV heart disease No history of active angina No myocardial infarction within 6 months No history of significant ventricular arrhythmia requiring medication No history of clinically significant conduction system abnormality Pulmonary: FEV1 at least 1.2 L Other: Not pregnant or nursing Negative pregnancy test No serious concurrent infections or uncontrolled nonmalignant medical illnesses No psychosis No clinically significant hearing loss No recurrent laryngeal nerve or phrenic nerve paralysis No concurrent active malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix Prior malignancies without evidence of disease for at least 5 years allowed

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy No other concurrent radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1997-08; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Bains MS, Stojadinovic A, Minsky B, Rusch V, Turnbull A, Korst R, Ginsberg R, Kelsen DP, Ilson DH. A phase II trial of preoperative combined-modality therapy for localized esophageal carcinoma: initial results. J Thorac Cardiovasc Surg. 2002 Aug;124(2):270-7. doi: 10.1067/mtc.2002.122545. PMID 12167786
- [Result] Enzinger E, Ilson D, Minsky B, et al.: Phase I/II neoadjuvant concurrent 96 hour taxol, cisplatin, and radiation therapy: promising toxicity profile and response in localized esophageal cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A1038, 1999.